CLINICAL TRIAL: NCT04337385
Title: The Effect of Prolonged vs. Interrupted Sitting With High Intensity Interval Exercise on Lower Limb Vascular Function in Adolescents Before and After a Mixed Meal
Brief Title: Interrupting Sitting With High Intensity Exercise on Vascular Function in Adolescents Before and After a Mixed Meal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 resulted in laboratory closures and the student has changed their research project in order to progress in their degree.
Sponsor: University of Exeter (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 191204/B/04
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Risk Factor; Endothelial Dysfunction
Keywords: Flow mediated dilation; Reactive hyperaemia; Endothelial function; Paediatrics; Physical inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 hours of Prolonged Sitting (Experimental): Participants will sit continuously for three hours before receiving a mixed meal challenge.
  Interventions: Behavioral: 3 hours of prolonged sitting
- 3 hours of interrupted sitting with hourly HIIE (Experimental): Participants will have their three hour sitting period interrupted with high intensity interval cycling exercise (HIIE) at 30, 90 and 150 minutes into the intervention. In each exercise bout, they will cycle at 90% peak power for 3 x 60 second periods with 75 seconds of recovery in-between.
  Interventions: Behavioral: Interrupting 3 hours of prolonged sitting with high intensity interval exercise

INTERVENTIONS:
Behavioral: Interrupting 3 hours of prolonged sitting with high intensity interval exercise — Breaking up a prolonged bout of sitting in adolescents using high intensity interval exercise
  Arms: 3 hours of interrupted sitting with hourly HIIE
Behavioral: 3 hours of prolonged sitting — Participants will be asked to remain seated for 3 hours and refrain from moving their lower limbs
  Arms: 3 hours of Prolonged Sitting

SUMMARY:
This study aims to investigate the effect of interrupting a three hour bout of prolonged sitting with high intensity interval exercise on lower limb blood vessel function in adolescents before and after a mixed meal challenge.

DETAILED DESCRIPTION:
Participants will be required to visit the laboratory on three separate occasions. The first of which will be a preliminary visit to collect anthropometric data (e.g. stature and body weight) and participants will complete a combined ramp-incremental and supra-maximal test to exhaustion on a cycle ergometer to determine the work rate for the exercise in the subsequent experimental visits.

For the two experimental visits, participants will arrive to the laboratory after an overnight fast and an activPAL accelerometer will be attached to the midline of the participants' thigh for the duration of the visit to quantity sitting time.

Lower limb macro and micro-vascular function will be assessed using a single protocol through flow mediated dilation of the popliteal artery and post-occlusive reactive hyperaemia in the capillaries of the calf. Participants will then either sit for three hours or have this three hour sitting period interrupted with high intensity interval cycling exercise at 30, 90 and 150 minutes. Vascular function will then be reassessed before participants will be given a mixed meal challenge (58.4 g fat and 53.4 g sugar) with a three hour postprandial period where the participants will remain seated for the duration. At the end of the postprandial period, vascular function will be reassessed.

Blood pressure, heart rate and calf circumference will be assessed hourly throughout the experimental day. In addition, capillary blood samples will be collected at baseline, pre meal and each hour during the postprandial period and assessed for changes in plasma glucose, triglyceride, cholesterol and insulin concentrations.

Participants will be transported to the toilet by wheelchair to limit the amount of walking undertaken during the sitting period and this activity will be quantified by the activPAL accelerometers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents
* 12-15 years

Exclusion Criteria:

* Medications known to affect blood pressure, carbohydrate or fat metabolism
* Allergies to the test meal e.g. dairy or gluten
* Contraindications to exercise
* Individuals with special educational needs that mean they are unable to fully comprehend the demands of the study procedures

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Popliteal macrovascular function | Before and after 3 hours of prolonged vs. interrupted sitting and after a subsequent 3 hour postprandial period
  Flow mediated dilation will be used to assess changes in microvascular function of the popliteal artery

SECONDARY OUTCOMES:
Microvascular function in the capillaries of the calf | Before and after 3 hours of prolonged vs. interrupted sitting and after a subsequent 3 hour postprandial period
  Microvascular function will be assessed using post occlusive reactive hyperaemia via laser Doppler flowmetry
Changes in plasma triglyceride concentration from a capillary sample | 6.5 hours
  Changes in plasma triglyceride concentration will be assessed in response to the prolonged or interrupted sitting and after mixed meal
Changes in plasma insulin concentration from a capillary sample | 6.5 hours
  Changes in plasma insulin concentration will be assessed in response to the prolonged or interrupted sitting and after mixed meal
Changes in plasma glucose concentration from a capillary sample | 6.5 hours
  Changes in plasma glucose concentration will be assessed in response to the prolonged or interrupted sitting and after mixed meal
Blood pressure | 6.5 hours
  Changes in blood pressure will be monitored hourly throughout the 3 hour sitting period and three hour postprandial period
Heart rate | 6.5 hours
  Changes in heart rate will be monitored hourly throughout the 3 hour sitting period and three hour postprandial period
Calf circumference | 6.5 hours
  Calf circumference will be monitored every hour throughout experimental visit to give an indication of venous pooling that may occur as a result of the prolonged sitting and be implicated in the potential decline in vascular function
Physical activity prior to the experimental visits | 48 hours prior to each visit
  Participants will wear GENEactiv accelerometers to monitor their physical activity levels before the experimental visit
Sitting time during the experimental visits | 6 hours
  Participants will wear an activPAL accelerometer on their thigh to quantify the amount of time they spend sitting, standing and cycling during the trials

OTHER OUTCOMES:
Participant Enjoyment During the High Intensity Interval Exercise | 3 hours
  The enjoyment of the high intensity interval exercise will be assessed during the exercise bouts using the Exercise Enjoyment Scale (ESS) (Stanley & Cumming, 2010). The scale runs from 1 (not at all) to 7 (extremely) so a larger score indicates greater enjoyment.
Participant Enjoyment Post the High Intensity Interval Exercise | 3 hours
  Participants will rate their enjoyment post exercise using the Physical Activity Enjoyment Scale (PACES) modified for adolescents (Motl et al., 2001). Participants rate how much they agree (1 = "disagree a lot" to 5 = "agree a lot") with 16 statements about their feelings from the exercise. The combined enjoyment scale score can range from 16 to 80 with a higher score indicating greater perceived enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Barker, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom